CLINICAL TRIAL: NCT02232464
Title: Disturbed Structural Connectivity of Frontostriatal and Frontoparietal Networks in Adults With Attention-deficit Hyperactivity Disorder
Brief Title: Disturbed Structural Connectivity of Frontostriatal and Frontoparietal Networks in Adults With ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201312144RINB
Record Dates: First submitted 2014-08-27; First posted 2014-09-05 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Adult ADHD; diffusion spectrum imaging; resting-state fMRI; frontostriatal circuitries; frontoparietal circuitries; executive function
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ADHD group: Adults with clinical diagnosis of ADHD according to the DSM-IV criteria
- Control group: Age-, sex-, and IQ-matched healthy controls without lifetime diagnosis with ADHD

SUMMARY:
Attention deficit/hyperactivity disorder (ADHD) is a common, impairing, childhood onset neuropsychiatric disorder with executive dysfunctions. The ADHD symptoms and executive deficits may last to adulthood. Our previous studies, like western results, have shown that children with ADHD have disrupted microstructural integrity of frontostriatal fiber pathways and impaired brain activity in frontoparietal network. However, there is lack of data with regards to whether adults with ADHD also demonstrate structural and functional disconnectivity of frontostriatal and frontoparietal networks as compared to healthy controls without ADHD in Asian population and no study has been done to correlate a wide range of executive functions with the connectivity of these two networks.

Specific Aims:

1. to compare the executive functions, and structural and functional connectivity in frontostriatal and frontoparietal circuitries between adults with ADHD and healthy controls without ADHD;
2. to correlate the data from structural and functional connectivity, executive functions, and ADHD core symptoms stratifying by the ADHD and controls; and
3. to explore other circuitries that may involve in ADHD by using whole brain tractography analyses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-45, who have clinical diagnosis of a ADHD according to the DSM-IV criteria.

Exclusion Criteria:

* The subjects will be excluded from the study if they meet any of the following criteria: (1) Comorbidity with diagnoses of autism spectrum disorder, schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorder, organic psychosis, schizotypal personality disorder, bipolar disorder, depression, severe anxiety disorders or substance use; (2) With neurodegenerative disorder, epilepsy, involuntary movement disorder, congenital metabolic disorder, brain tumor, history of severe head trauma, and history of craniotomy; (3)With visual or hearing impairments, or motor disability which may influence the process of MRI assessment; and (4) Full-scale IQ lower than 80.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample consists of 50 adults (ages 18-45) with clinical diagnosis of ADHD according to the DSM-IV criteria and 50 age-, sex-, and IQ-matched healthy controls without lifetime diagnosis with ADHD.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Structural neuroimaging | one day
  Using diffusing spectrum imaging (DSI) to assess the structural connectivity in frontostriatal, frontoparietal and other circuitries.

SECONDARY OUTCOMES:
Functional connectivity of the brain circuits | one day
  Using resting-state functional MRI (rsfMRI) to assess the functional connectivity in frontostriatal, frontoparietal and other circuitries.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan